CLINICAL TRIAL: NCT02465294
Title: The Influence of Probiotics With a Behavioral Life Style Intervention on Body Weight and Composition in Overweight Participants: A Randomized, Double-blinded, Placebo-controlled Study.
Brief Title: The Influence of Probiotics on Body Weight and Composition
Acronym: WLP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study withdrawn due to funding
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201400484
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Healthy; Overweight
Keywords: Probiotics; Weight loss; Body composition
MeSH Terms: conditions — Overweight; Weight Loss | interventions — Probiotics; Lacteol; stearic acid; Hematologic Tests

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Potato starch and magnesium stearate (Placebo Comparator): This arm will be used as a control to asses the efficacy of the other probiotic arms. The placebo will contain encapsulated potato starch and magnesium stearate which is used the matrix in the probiotic supplements. The placebo refers only to the intervention supplement, not the behavioral lifestyle intervention. All subjects will participate in the same behavioral lifestyle intervention. In addition, blood tests will be performed.
  Interventions: Behavioral: Behavioral lifestyle intervention; Other: Placebo; Other: Blood Test
- Lactobacillus (Experimental): Lactobacillus will be taken as a capsule once daily for 12 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded). All subjects will participate in the same behavioral lifestyle intervention. In addition, blood tests will be performed.
  Interventions: Dietary Supplement: Probiotic; Behavioral: Behavioral lifestyle intervention; Other: Blood Test
- Mix of Bifidobacterium and Lactobacillus (Experimental): A blend of Bifidobacterium and Lactobacillus will be taken as a capsule once daily for 12 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded). All subjects will participate in the same behavioral lifestyle intervention. In addition, blood tests will be performed.
  Interventions: Behavioral: Behavioral lifestyle intervention; Other: Blood Test; Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — This group will receive the Lactobacillus probiotic, which will be taken as a capsule once daily for 12 weeks.
  Other Names: Lactobacillus
  Arms: Lactobacillus
Behavioral: Behavioral lifestyle intervention — All participants will participate in weekly group meetings of 15 to 20 participants for a facilitated discussion of specific nutritional, behavioral, and physical activity topics chosen to promote weight loss.
Other: Placebo — This group will receive the placebo and will be taken as a capsule once daily for 12 weeks. The placebo will contain encapsulated potato starch which is used the matrix in the probiotic supplements.
  Other Names: Potato starch and magnesium stearate
  Arms: Potato starch and magnesium stearate
Other: Blood Test — All subjects will have blood tests performed.
Dietary Supplement: Probiotic — This group will receive the blend of Bifidobacterium and Lactobacillus probiotic, which will be taken as a capsule once daily for 12 weeks.
  Other Names: A blend of Bifidobacterium and Lactobacillus
  Arms: Mix of Bifidobacterium and Lactobacillus

SUMMARY:
The purpose of this study is to evaluate the addition of two different probiotic interventions to a comprehensive behavioral lifestyle intervention on body weight loss and overall health in overweight adults.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled study. After obtaining informed consent, healthy overweight adults aged 18 to 75 years (n=76/intervention group with n=228 total/study) will be randomized to one of three groups: Lactobacillus, a blend of Bifidobacterium and Lactobacillus, or placebo. Participants will consume 1 capsule per day of probiotic or placebo for 12 weeks. Participants will attend weekly behavioral lifestyle intervention meetings, which will address dietary and physical activity contributions to weight loss, in groups of approximately 20 subjects during the 12 intervention weeks.

Participants will complete daily questionnaires throughout the week before and during the intervention period which address subject compliance and bowel habits. A dual X-ray absorptivity scan will be done to measure body composition during the week before the intervention and during the 12th week of the intervention period (± 1 week). Blood samples will be collected via a finger prick at the baseline and final time points. Blood samples will be used to measure cardiovascular and metabolic markers of health. Stool samples will be collected from 25 subjects per intervention group during the week before the intervention period and the 12th week of the intervention period. Dietary intake will be assessed during the week before the intervention period and during the week of the final appointment (± 1 week). Gastrointestinal symptoms and physical activity questionnaires will be completed upon providing consent to the study, being randomized to an intervention, and during the last week of the intervention period. Questionnaires regarding income, weight control strategies, and quality of life will be completed during randomization and during the last week of the intervention period. Stool samples will be collected from a subgroup of participants during the week before the intervention period and during the 12th week of the intervention period. These samples will be used to detect the presence and/or abundance and/or survival of the probiotic microorganisms at the end of the digestive tract.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study you must:

* Be age 18 to 75 years
* Have a BMI ≥ 25
* Be willing to receive random assignment to probiotic or placebo supplementation
* Be willing to and able to complete the Informed Consent Form in English
* Be willing to complete questionnaires, records, and diaries associated with the study and to complete all study visits
* Be committed to losing weight over the 12-week study period
* Be willing to discontinue consumption of fermented foods or probiotics (e.g., yogurts with live, active cultures or supplements).
* Be willing to provide a social security number (SS#) to receive study payment? Note: the subject can still participate if unwilling to provide SS#, but no financial reimbursement can be provided.

Exclusion Criteria:

To participate in the study you must NOT:

* Have used another investigational product within 3 months of enrolling in the study
* Be pregnant or breast-feeding or planning on becoming pregnant in the next 18 months
* Be allergic to milk, soy, or yeast
* Have gained or lost at least 10 lbs in the previous 3 months
* Have had uncontrolled angina (severe chest pain) within the past 6 months
* Have insulin-dependent diabetes (oral medications are not exclusionary)
* Use weight-loss medications
* Have had cancer treatment (radiation, chemotherapy, or surgery) within the past 6 months or any other treatment or condition known to weaken the immune system (e.g., systemic corticosteroids or HIV/AIDS)
* Be currently being treated for or have any of the following physician-diagnosed diseases or conditions: inflammatory bowel disease, celiac disease, short bowel syndrome, or any other malabsorptive syndrome?
* Have any physical condition deemed likely to significantly interfere with your ability to participate in a lifestyle intervention involving eating and physical activity changes
* Be currently participating in Weight Watcher's or another weight loss program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Changes in baseline to week 12 in the percentage of body weight lost between the probiotic groups and the placebo group | Change from Baseline (start of week 1) to Week 12
  Body weight (kg)

SECONDARY OUTCOMES:
Changes in body composition (Fat mass) between the probiotic groups and the placebo group | Changes from Pre-baseline to Week 12
  Fat mass (kg)
Changes in body composition (Waist circumference) between the probiotic groups and the placebo group | Changes from Pre-baseline to Week 12
  Waist circumference (cm)
Changes in body composition (Sagittal abdominal diameter) between the probiotic groups and the placebo group | Changes from Pre-baseline to Week 12
  Sagittal abdominal diameter (cm)
Changes in bowel habits between the probiotic groups and the placebo group | Changes from Pre-baseline (Week -1) to Week 12
  Bowel movement frequency (average number per week)
Changes in gastrointestinal symptoms between the probiotic groups and the placebo group | Changes from Pre-baseline (Week -1) to Week 12
  Symptoms measured using the Gastrointestinal Symptom Rating Score questionnaire provide a score for the follow five syndromes: abdominal pain, reflux, constipation, diarrhea, and indigestion.
Changes in markers of cardiovascular health between the probiotic groups and the placebo group | Changes from Pre-baseline to Week 12
  Serum cholesterol (mg/dl)
Changes in nutritional intake between the probiotic groups and the placebo group | Changes from Pre-baseline (Week -1) to Week 12
  Total energy intake (kcal) will be assessed using the automated self-administered 24 hour dietary recall.
Changes in weight control strategies between the probiotic groups and the placebo group | Changes from Pre-baseline (Week -1) to Week 12
  Differences in weight control strategies questionnaire scores
Changes in intestinal microbiota community composition between the probiotic groups and the placebo group | Changes from Pre-baseline (Week -1) to Week 12
  Stool samples will be collected from a subgroup of participants to analyze intestinal microbiota community composition.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No